CLINICAL TRIAL: NCT05044988
Title: A Single-arm, Open-label, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of HS-10342 in Previously Treated Patients With Hormone Receptor Positive and Human Epidermal Growth Factor Receptor 2 Negative Advanced and/or Metastatic Breast Cancer
Brief Title: A Study of HS-10342 in Chinese Patients With HR+/HER2- Advanced and/or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10342-201
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: HR+/HER2- Advanced and/or Metastatic Breast Cancer
Keywords: Advanced and/or Metastatic Breast Cancer; HR+/HER2-; CDK4/6; HS-10342

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10342 (Experimental): Each subject will receive repeat doses (C1, C2…) for 28-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: HS-10342

INTERVENTIONS:
Drug: HS-10342 — HS-10342 tablet once daily from Day 1 to 21 of a 28-day cycle

SUMMARY:
HS-10342 is a selective CDK4/6 kinase inhibitor. This study is conducted to evaluate the safety and efficacy of HS-10342 at repeated doses.

DETAILED DESCRIPTION:
HS-10342-201 is a single- arm, open- label, multicenter, phase 2 study in patients with hormone receptor positive (HR positive), human epidermal growth factor receptor 2 negative (HER2 negative) advanced and/or metastatic breast cancer who have had disease progression after endocrine therapy. The efficacy is evaluated as monotherapy, and the primary endpoint is ORR.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of Hormone Receptor Positive(HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) breast cancer.
2. Recurrent, locally advanced, unresectable or metastatic breast cancer with disease progression following anti-estrogen therapy.
3. Prior treatment with chemotherapy regimens, No more than 2 prior chemotherapy regimens in the metastatic setting.
4. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
5. recovered from the acute effects of therapy with toxicity resolving to baseline or grade 1 except for residual alopecia and peripheral neuropathy.
6. Adequate function of major organs.

Exclusion Criteria:

1. Has received or is undergoing the following treatments:

   1. Currently receiving or have received any CDK4/6 inhibitors;
   2. Receiving/received antitumor therapy within 14 days or 5 half-lives, before the initial dose whichever is the longer;
   3. Radiotherapy with a limited field of radiation for palliation within 14 days of the initial dose of study drug, or received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 28 days of the initial dose.;
   4. Major surgery within 4 weeks of the initial dose of study drug;
   5. Brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study treatment. Meningeal or brainstem metastases. Spinal cord compression;
2. Abnormal liver and kidney functions that are known to affect drug metabolism and excretion:
3. History of other primary malignancies.
4. Participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Complete Response (CR) or Partial Response (PR)（Objective response rate [ORR]） | Up to approximately 12 months
  ORR was the percentage of participants achieving a best overall response (BOR) of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions.

SECONDARY OUTCOMES:
Overall Survival (OS) | From Date of the First Dose until Death Due to Any Cause (Up To 24 Months)
  OS defined as the time from first dose date to the date of death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Duration of Response (DOR) | From Date of CR, PR until Disease Progression or Death Due to Any Cause (Up To 12 Months)
  DOR was the time from the date of first evidence of CR or PR to the date of objective progression or the date of death due to any cause, whichever is earlier.
Progression Free Survival (PFS) | From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 24 Months)
  PFS defined as the time from the first day of therapy to the first evidence of disease progression as defined by RECIST v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of first dose, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Percentage of Participants With CR, PR or SD | Disease Control Rate [DCR]) [ Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up To 12 Months)
  Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions.